CLINICAL TRIAL: NCT01636609
Title: Phase I/II Study of Cytarabine or 5-Azacitidine Combined With Tosedostat to Evaluate the Safety and Tolerability in Older Patients With Acute Myeloid Leukemia (AML) or High Risk MDS
Brief Title: Tosedostat and Cytarabine or Azacitidine in Treating Older Participants With Acute Myeloid Leukemia or High Risk Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: In 2013 the FDA put a temporary hold on the trial and the Phase II portion of this study was cancelled.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0188; NCI-2018-01817 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2011-0188 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Acute Myeloid Leukemia; High Risk Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Cytarabine; tosedostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (tosedostat, cytarabine) (Experimental): Participants receive tosedostat PO QD on days 1-28 and cytarabine SC BID on days 1-10. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Drug: Tosedostat
- Arm II (tosedostat, azacitidine) (Experimental): Participants receive tosedostat PO QD on days 1-28 and azacitidine IV over 10-40 minutes or SC on days 1-7. Courses repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Tosedostat

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: Arm II (tosedostat, azacitidine)
Drug: Cytarabine — Given SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Arm I (tosedostat, cytarabine)
Drug: Tosedostat — Given PO
  Other Names: Aminopeptidase inhibitor CHR-2797; CHR-2797

SUMMARY:
This phase I/II trial studies the side effects and best dose of cytarabine and azacitidine and how well they work when giving together with tosedostat in treating older participants with acute myeloid leukemia or high risk myelodysplastic syndrome. Tosedostat and azacitidine may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving tosedostat and cytarabine or azacitidine may work better in treating participants with acute myeloid leukemia or high risk myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety profile of tosedostat (oral) in combination with cytarabine (subcutaneous [SQ]) or azacitidine (5-azacytidine) in patients age 60 years or older with relapsed/refractory acute myeloid leukemia (AML) or high risk myelodysplastic syndrome (MDS).

II. To observe the anti-tumor effects of tosedostat in combination with cytarabine or 5-azacytidine, if any occur.

OUTLINE: This is a phase I, dose-escalation of cytarabine and azacitidine followed by a phase II study. Participants are assigned to 1 of 2 arms.

ARM I: Participants receive tosedostat orally (PO) once daily (QD) on days 1-28 and cytarabine subcutaneously (SC) twice daily (BID) on days 1-10. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Participants receive tosedostat PO QD on days 1-28 and azacitidine intravenously (IV) over 10-40 minutes or SC for on days 1-7. Courses repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants will be followed up at 28 days and then every 3-5 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Signed, informed consent must be obtained prior to any study specific procedures
* For the phase I portion of the study patients should have failed any number of prior therapies, which should include at least the following:

  * Patients with MDS should have failed prior therapy with a hypomethylating agent and/or with lenalidomide
  * Patients with AML should have failed any prior induction therapy or have relapsed after prior therapy
  * Patients with MDS who received therapy with a hypomethylating agent and progress to AML are eligible at the time of diagnosis of AML regardless of any prior therapy for AML
  * Patients with any of the eligible diagnoses who have received no prior therapy are eligible if not candidates to receive standard therapy or if they refuse standard chemotherapy
* For the phase II portion of the study, only patients who are previously untreated for AML. 1. Patients with history of MDS who received therapy for MDS and progressed to AML are eligible at the time of diagnosis of AML. Only induction chemotherapy administered for AML will be considered for considerations of eligibility regarding prior therapy. Patients who received therapy for MDS before transforming to AML (e.g., with hypomethylating agents or lenalidomide) are eligible
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use acceptable contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) while on study and must continue to do so for 3 months after stopping study drug, and must have a negative urine or serum pregnancy test within 2 weeks prior to beginning treatment on this trial. Sexually active men must also use acceptable contraceptive methods for the duration of time on study. Pregnant and nursing patients are excluded because the effects of tosedostat on a fetus or nursing child are unknown
* Patients must have been off chemotherapy for 2 weeks prior to entering this study, unless there is evidence of rapidly progressive disease, and must have recovered from the toxic effects of that therapy to at least grade 1. Use of hydroxyurea for patients with rapidly proliferative disease is allowed before the start of study therapy and for the first four weeks on therapy
* Serum creatinine =< 2.0 mg/dl
* Total bilirubin =< 1.5 x the upper limit of normal unless considered due to Gilbert's syndrome
* Alanine aminotransferase (ALT), or aspartate aminotransferase (AST) =< 3 x the upper limit of normal
* Left ventricular ejection fraction (LVEF) >= 50% within 28 days prior to first dose of study drug administration
* Patient is able to comply with all study procedures including study drug administration, visits and tests
* For patients with history of anthracycline exposure or coronary artery disease co-management by cardiology to optimize cardioprotective medications will be required prior to tosedostat initiation

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to uncontrolled infection, symptomatic congestive heart failure (New York Heart Association class III or IV), or psychiatric illness/social situations that would limit compliance with study requirements
* Active heart disease including myocardial infarction within previous 6 months, symptomatic coronary artery disease, clinically significant arrhythmias not controlled by medication, atrial fibrillation (whether active or known past history), uncontrolled angina, or uncontrolled congestive heart failure (New York Heart Association class III or IV)
* Recent exposure to cardiotoxic agents (including anthracyclines) within 3 months of enrollment. Subjects with troponin-I and brain natriuretic peptide (BNP) levels above upper limit of normal (ULN) are excluded
* Patients with acute promyelocytic leukemia (APL) (FAB type M3) or chronic myelogenous leukemia (CML) in blast crisis
* Significant gastrointestinal disorders that may interfere with absorption of tosedostat
* Patients who have received a stem cell transplant in the past
* Patients who can receive an allogeneic stem cell transplant within 4 weeks
* Use of concomitant drugs that prolong QT/corrected QT (QTc) interval are prohibited with the exception of antibiotics, antifungals, and other antimicrobials that are used as standard of care to prevent or treat infections and other such drugs that are considered absolutely essential for the care of the patient, but only if clinically indicated and must be fully documented

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-11-20 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of cytarabine and azacitidine (Phase I) | Up to 28 days
Overall response defined as complete response (CR), CR with incomplete platelet recovery (CRp) or CR with insufficient hematological recovery (CRi), morphologic leukemia free state (MLF), partial response (PR), or hematologic improvement (HI) | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org